CLINICAL TRIAL: NCT04842058
Title: Pathophysiologic Hemodynamics After Primary Unilateral Total Hip Arthroplasty in Patients Receiving Angiotensin-Converting Enzyme Inhibitors (ACEIs) and Angiotensin II Receptor Blockers (ARBs)
Brief Title: Pathophysiologic Hemodynamics After Primary Unilateral Total Hip Arthroplasty in Patients Receiving ACEIs and ARBs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hvidovre University Hospital (Other)
Collaborators: Kehlet, Henrik, M.D., Ph.D. (Individual)
Responsible Party: Principal Investigator, Ana-Marija Hristovska, MD, Hvidovre University Hospital
Other Study IDs: H-20017723
Record Dates: First submitted 2021-04-08; First posted 2021-04-12 (Actual); Last update posted 2021-04-12 (Actual); Status verified 2021-04

CONDITIONS: Orthostatic Intolerance; Orthostatic Hypotension
Keywords: Orthostatic Hypotension; Orthostatic Intolerance; Postoperative period; Antihypertensives; Autonomic dysfunction
MeSH Terms: conditions — Orthostatic Intolerance; Hypotension, Orthostatic; Primary Dysautonomias

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orthostatic tolerant patients (OT): Patients that experience symptoms of orthostatic intolerance (dizziness, nausea, vomiting, blurry vision or syncope) or orthostatic hypotension (fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg) during mobilisation
  Interventions: Other: Mobilisation procedure
- Orthostatic intolerant patients (OI): Patients that do not experience symptoms of orthostatic intolerance (dizziness, nausea, vomiting, blurry vision or syncope) or orthostatic hypotension (fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg) during mobilisation
  Interventions: Other: Mobilisation procedure

INTERVENTIONS:
Other: Mobilisation procedure — A standardized mobilization procedure was performed preoperatively ~ 1h before surgery and was repeated 6h and 24h after surgery. The mobilization procedure included patient supine rest (5 minutes), followed by 45° passive leg raise (PLR) (3 minutes), supine rest (5 minutes), sitting on the edge of the bed with feet resting on the floor (3 minutes) followed by standing using a walker while the patient was encouraged verbally to stand on toes and shift body weight from one leg to the other (3 minutes) and finally rest in supine position (5 minutes). The procedure was terminated prematurely in any position if patients experienced unbearable symptoms of OI or upon a decrease of systolic arterial pressure (SAP) > 30 mmHg.

SUMMARY:
Incidence and pathophysiologic hemodynamics of postoperative orthostatic intolerance and orthostatic hypotension in patients receiving antihypertensives

DETAILED DESCRIPTION:
Early postoperative mobilization is essential for rapid functional recovery after surgery and it is considered a cornerstone in the so-called fast track multimodal perioperative approach, which includes early ambulation, oral nutrition, multimodal opioid-sparing analgesia and optimized fluid therapy. This strategy has improved patient outcome after surgery and reduced hospital length of stay. Immobilization after surgery is associated with increased risk of complications including venous thromboembolism (deep venous thrombosis, pulmonary embolism), muscle wasting, pneumonia and atelectasis, thereby impending convalescence.

However, early postoperative mobilization can be delayed due to failed orthostatic cardiovascular regulation, resulting in postoperative orthostatic hypotension (OH), defined as a decrease in systolic blood pressure > 20 mmHg or diastolic blood pressure > 10 mmHg or postoperative orthostatic intolerance (OI), characterized by dizziness, nausea, vomiting, visual disturbances or syncope.

Previous studies investigating the incidence and pathophysiology of postoperative OI and OH included mixed patient populations. Hitherto no studies have been performed looking into the incidence and pathophysiologic hemodynamics of postoperative OI and OH specifically in patients receiving angiotensin-converting enzyme inhibitors (ACEIs) and angiotensin II receptor blockers (ARBs), antihypertensive agents with potential effects on cardiovascular compensatory functions.

The current study aims therefore to estimate the incidence and gain knowledge on pathophysiological hemodynamics of postoperative OI and OH in patients receiving ACEIs and ARBs.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary unilateral total hip arthroplasty (THA) in spinal anaesthesia in standardized fast-track setting
* Habitual use of angiontensin-Converting Enzyme Inhibitors (ACEIs) and/or angiotensin 2 receptor blockers (ARBs) on any indication
* Patients > 18
* Patients that understand and speak Danish
* Patients that have provided written informed consent

Exclusion Criteria:

* Alcohol abuse
* Any type of substance abuse
* Chronic pain treated by habitual use of opioids
* Habitual use of anxiolytic, antidepressant and/or antipsychotic drugs
* History of cerebral apoplexy or transitory cerebral ischemia
* History of previous orthostatic intolerance or hypotension
* History of diabetes mellitus
* History of following diseases of the autonomic nervous system: Parkinson disease, multiple sclerosis, multiple system atrophy, autonomic neuropathies
* Cognitive dysfunction
* Dementia
* American Society of Anesthesiologists (ASA) > 3

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients receiving antuhypertensives (ACEIs, ARBs) and undergoing primary unilateral total hip arthroplasty in spinal anesthesia in standardized fast-track setting
Sampling Method: Probability Sample
Enrollment: 24 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of orthostatic intolerance | 6 hours postoperatively
  Symptoms of orthostatic intolerance: dizziness, nausea, vomiting, blurry vision or syncope during mobilization
Incidence of orthostatic hypotension | 6 hours postoperatively
  Orthostatic hypotension is defined as a fall in systolic pressure > 20 mmHg and/or diastolic pressure > 10 mmHg during mobilization

SECONDARY OUTCOMES:
Changes in systolic arterial pressure (SAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg by non-invasive Lithium Dilution Cardiac Output (LiDCO) measurement
Changes in diastolic arterial pressure (DAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg by non-invasive LiDCO
Changes in mean arterial pressure (MAP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg by non-invasive LiDCO
Changes in systemic vascular resistance (SVR) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in dynes s cm-5 by non-invasive LiDCO
Changes in cardiac output (CO) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in L/min by non-invasive LiDCO
Changes in stroke volume (SV) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL by non-invasive LiDCO
Changes in heart rate (HR) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in beats min-1 by non-invasive LiDCO
Changes in pulse pressure (PP) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in mmHg
Changes in cerebral perfusion (ScO2) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in % by Root Masimo
Changes in muscular perfusion (SmO2) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in % by Root Masimo
Changes in peripheral perfusion index (PPI) during mobilization | Preoperatively, 6 and 24 hours postoperatively
  Measured in % by Root Masimo
Changes in total blood volume (TBV) | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL by Carbon Monoxide - rebreathing technique
Changes in red blood cell volume (RBCV) | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL by Carbon Monoxide - rebreathing technique
Changes in plasma volume (PV) | Preoperatively, 6 and 24 hours postoperatively
  Measured in mL by Carbon Monoxide - rebreathing technique
Changes in hematocrit | Preoperatively, 6 and 24 hours postoperatively
  Measured in %
Changes in total mass of hemoglobin | Preoperatively, 6 and 24 hours postoperatively
  Measured in grams
Changes in hemoglobin concentration | Preoperatively, 6 and 24 hours postoperatively
  Measured in gr/L
Changes in C-Reactive Protein | Preoperatively, 6 and 24 hours postoperatively
  Measured in mg/L
Changes in heart rate variability (HRV) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured in ms
Changes in baroreflex sensitivity - vagal (BRSv) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured in ms
Changes in Valsalva ratio (VR) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured as index
Changes in Systolic Sympathetic Index 1 (SSI1) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured as index
Changes in Systolic Sympathetic Index 2 (SSI2) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured as index
Changes in Systolic Sympathetic Index 3 (SSI3) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured as index
Changes in Diastolic Sympathetic Index 1 (DSI1) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured as index
Changes in Diastolic Sympathetic Index 2 (DSI2) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured as index
Changes in Diastolic Sympathetic Index 3 (DSI3) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured as index
Changes in Pressure Recovery Time (PRT) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured in seconds
Changes in Baroreceptor Reflex Sensitivity-adrenergic (BRS-a) during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured in seconds
Changes in systolic latency during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured in seconds
Changes in diastolic latency during Valsalva manoeuvre | Preoperatively, 6 and 24 hours postoperatively
  Measured in seconds

OTHER OUTCOMES:
Pain score during mobilisation | Preoperatively, 6 and 24 hours postoperatively
  Measured by verbal rating scale (VRS) from 0 to 10 (0 = no pain, 10 = worse pain imaginable)
Estimated intraoperative bleeding | During surgery
  Measured in mL
Intraoperative fluid balance | Intraoperative
  Measured in mL
Surgery duration | Intraoperative
  Minutes
Intraoperative propofol usage | Intraoperative
  Mg
Usage of cumulated opioids prior to mobilisation | Postoperatively
  mg
Usage of Chlorzoxazone prior to mobilisation | Postoperatively
  mg
Preoperative use of antihypertensives | Preoperatively
  Type, dose and time of administration
Postoperative use of antihypertensives | Postoperatively
  Type, dose and time of administration

CONTACTS AND LOCATIONS:
Locations (1):
- Hvidovre University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Jans O, Bundgaard-Nielsen M, Solgaard S, Johansson PI, Kehlet H. Orthostatic intolerance during early mobilization after fast-track hip arthroplasty. Br J Anaesth. 2012 Mar;108(3):436-43. doi: 10.1093/bja/aer403. Epub 2011 Dec 15. PMID 22174345
- [Background] Jans O, Kehlet H. Postoperative orthostatic intolerance: a common perioperative problem with few available solutions. Can J Anaesth. 2017 Jan;64(1):10-15. doi: 10.1007/s12630-016-0734-7. Epub 2016 Sep 14. No abstract available. PMID 27638295